CLINICAL TRIAL: NCT05556538
Title: The Effect of Subcutaneous Fat Tissue Thickness on Lumbar Transforaminal Epidural Steroid Injection Treatment Success
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-AS-SŞ-22.09.22
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Disc Herniation; Radiculopathy Lumbar; Obesity
Keywords: Transforaminal Epidural Injection; Subcutaneous Fat Tissue Thickness; Subcutaneous Fat Index; Lumbar Disc Hernia; Radicular Pain; Obesity
MeSH Terms: conditions — Intervertebral Disc Displacement; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Those who had TFESI and whose subcutaneous fat index was above the cut-off value: Those who are above the subcutaneous fat index cut-off values (9.4 mm in men, 8.45 mm in women) will be included in this group.
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- Those who had TFESI and whose subcutaneous fat index was below the cut-off value: Those who are below the subcutaneous fat index cut-off values (9.4 mm in men, 8.45 mm in women) will be included in this group.
  Interventions: Procedure: Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: Transforaminal Epidural Steroid Injection — Patients are placed in the prone position, with a pillow under their abdomen (to reduce lumbar lordosis) and taken to the operating table. The procedure area is cleaned 3 times with povidone-iodine antiseptic and covered with a sterile cover. In order to view the foramen to be processed, the fluoroscopy arm is evaluated at AP-oblique / cranial or caudal angles to obtain an optimal image. Local anesthetic (3 cc 2% prilocaine) is injected into the skin and subcutaneous tissue. The spinal Quincke 21-gauge 90 mm needle is advanced by targeting the relevant foramen under the guidance of fluoroscopy image. Needle position is confirmed by taking a lateral view. Needle aspiration is checked for blood. 1-2 ml of contrast material is injected to confirm that there is no vascular distribution and that it is in the epidural space. When distribution without vascular invasion is observed, an injection of a mixture of 10 mg dexamethasone, 1 cc saline and 1 cc (0.5%) bupivacaine is performed.

SUMMARY:
Nerve compression due to lumbar disc herniation and related radicular pain is a very common condition when the lifetime prevalence is considered. Lumbosacral radicular pain can be defined as pain originating from the lumbar level and spreading to the lower extremities along the distribution area of one or more spinal nerves. It is thought that the mechanical pressure of the disc material herniated to the dorsal nerve root or ganglion or the inflammation created by the chemokines and enzymes in the disc are involved in the pain formation mechanism.

Various methods such as medical agents, physical therapy modalities, epidural steroid injections and surgical methods can be used in the treatment of the related condition. Epidural injections have been used for the treatment of lower back and lower extremity pain since about 1900. Epidural injections exert their effects through the anti-inflammatory and neural membrane stabilizing effects of steroids, as well as by local anesthetics increasing blood flow to the ischemic spinal root and by the removal of cytokines from the area by the injection material. Epidural injections can be performed with various different approaches, including caudal, interlaminar and transforaminal. Among these approaches, the transforaminal approach is the most recently developed approach in the late 1990s, which allows drugs to be administered directly to the pathology area.

The effect of obesity, which is one of the factors thought to predispose to low back pain and lumbosacral radicular pain, has been evaluated in various studies and it has been found that it is positively correlated with low back pain and is an independent risk factor for lumbar herniation. So, does obesity have an effect on the success of transforaminal epidural steroid injection treatment? According to the literature, no significant effect on treatment success has been demonstrated.

Although the body mass index, which is used in the evaluation of obesity, has provided us important information about the health of the person in general for a long time, it is now thought to lead to an incomplete assessment. Because it does not provide information about body composition ratios (fat amount / lean body mass). Studies have shown that there is a high correlation between the percentage of body fat and the thickness of the subcutaneous fat tissue in the lumbar region, and there is a significant relationship between the lumbar region subcutaneous fat tissue thickness (especially L1-L2 level) and the degree of intervertebral disc degeneration and vertebral surface change. From this point of view, in another study, the L1-L2 disc level subcutaneous fat tissue thickness, was called the subcutaneous fat index, and the cut-off values that showed a significant relationship with spinal degeneration were determined.

In the study we planned, in cases of spinal radicular pain (etiologically caused by intervertebral disc herniation), body mass index, lumbar level subcutaneous fat tissue thickness and subcutaneous fat index data whether be or be not correlated with treatment effectiveness/success in patients who received transforaminal epidural steroid injection, and if so, the level of significance intended to work. Before applying for surgery, we aim to develop a practical approach that can be used by relevant clinicians and contribute to the literature, which can predict 'what level of treatment success can we achieve in which patient?' with this injection method.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Patients with a diagnosis of lumbosacral radiculopathy with low back and leg pain for at least 3 months that did not respond to other treatment methods
* Çalışmaya katılma için gönüllü olmak ve onam formu imzalamış olmak
* Presence of single root nerve compression due to MR imaging-proven single-level lumbar disc herniation
* Completeness of 3-month clinical evaluation data after the procedure

Exclusion Criteria:

* Having had lumbosacral surgery
* Multilevel disc herniation
* Presence of foraminal disc herniation
* Presence of local and/or systemic infection
* History of malignancy
* Presence of spinal stenosis
* Pregnancy
* Presence of known coagulopathy
* Having a known psychiatric illness diagnosis
* History of allergy to any of the injection substances
* Epidural steroid injection in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will consist of patients who are planned to receive transforaminal epidural steroid injection treatment by the clinician, and who want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Treatment Success | 3 weeks after TFESI
  More than 50% reduction in NRS (Numeric Rating Scale) and more than 40% reduction in ODI (Oswestry Disability Index) will be taken as criteria.
  (NRS is a scale that is defined as '0' = no pain, '10' = the most severe, unbearable pain, in which the patient gives points between '0' and '10' for the low back and leg pain felt by the patient.)
  (ODI is a deficiency/competence index that includes assessments grouped according to the types of daily activities in patients with low back pain.)
Treatment Success | 3 months after TFESI
  More than 50% reduction in NRS (Numeric Rating Scale) and more than 40% reduction in ODI (Oswestry Disability Index) will be taken as criteria.
  (NRS is a scale that is defined as '0' = no pain, '10' = the most severe, unbearable pain, in which the patient gives points between '0' and '10' for the low back and leg pain felt by the patient.)
  (ODI is a deficiency/competence index that includes assessments grouped according to the types of daily activities in patients with low back pain.)

SECONDARY OUTCOMES:
NRS (Numeric Rating Scale) | Before TFESI / 1 Hour After TFESI / 3 weeks after TFESI / 3 months after TFESI
  NRS is a scale that is defined as '0' = no pain, '10' = the most severe, unbearable pain, in which the patient gives points between '0' and '10' for the low back and leg pain felt by the patient.
ODI (Oswestry Disability Index) | Before TFESI / 3 weeks after TFESI / 3 months after TFESI
  ODI is a deficiency/competence index that includes assessments grouped according to the types of daily activities in patients with low back pain.
SF-12 (12-item Short Form Survey) | Before TFESI / 3 weeks after TFESI / 3 months after TFESI
  SF-12 is a scale that evaluates the patient's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No